CLINICAL TRIAL: NCT02062827
Title: A Phase 1 Study of M032 (NSC 733972), a Genetically Engineered HSV-1 Expressing IL-12, in Patients With Recurrent/Progressive Glioblastoma Multiforme, Anaplastic Astrocytoma, or Gliosarcoma
Brief Title: Genetically Engineered HSV-1 Phase 1 Study for the Treatment of Recurrent Malignant Glioma
Acronym: M032-HSV-1
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, James Markert, MD, Principal Investigator, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UAB-1317; R01CA217179 (NIH)
Record Dates: First submitted 2014-02-09; First posted 2014-02-14 (Estimated); Results first posted 2024-02-02 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Recurrent Glioblastoma Multiforme; Progressive Glioblastoma Multiforme; Anaplastic Astrocytoma or Gliosarcoma
Keywords: Glioma; Virus; Oncolytic virus; Gene therapy; Immunotherapy; Brain Tumors
MeSH Terms: conditions — Glioblastoma; Astrocytoma; Gliosarcoma; Glioma; Virus Diseases; Brain Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Group A single dose of HSV-1 (M032) (Experimental): single dose of HSV-1 (M032) infused through catheters into region(s) of tumor defined by MRI
  Interventions: Biological: M032 (NSC 733972)

INTERVENTIONS:
Biological: M032 (NSC 733972) — A single dose of HSV-1 (M032) infused through catheters into region(s) of tumor defined by MRI

SUMMARY:
To determine the safety and tolerability of the maximum dose for laboratory engineered Herpes Simplex Virus-1 in patients who would not be eligible for surgical resection of recurrent glioma To determine the safety and tolerability of the maximum dose for laboratory engineered Herpes Simples Virus-1 in patients who would benefit from surgical resection of recurrent glioma

DETAILED DESCRIPTION:
M032 is a second-generation oncolytic herpes simplex virus (oHSV) that is conditionally replication competent; that is, similar to G207, a first generation oHSV, it can replicate in tumor cells, but not in normal cells, thus killing the tumor cells directly through this process. Replication of M032 in the tumor itself not only kills the infected tumor cells, but causes the tumor cell to act as a factory to produce new virus. These virus particles are released as the tumor cell dies, and can then proceed to infect other tumor cells in the vicinity, and continue the process of tumor kill. In addition to this direct oncolytic activity, the virus carries a therapeutic payload--acting as a gene therapy vector, too--and causes the tumor cell to synthesize and secrete an immunity-stimulating protein called Interleukin-12 (IL-12) before it is killed. This IL-12 is released and promotes an immune response against surviving tumor cells, which increases the antitumor effect of the therapy. The IL-12 that is expressed can also produce an anti-angiogenic effect, by interfering with the production of new tumor blood vessels necessary to allow tumor growth. Anti-angiogenic therapies potentially starve the tumor of necessary oxygen and nutrients. Thus, the M032 oHSV produces three different potential mechanisms for antitumor effects. The virus has also been genetically-engineered to minimize the production of any toxic effects for the patient receiving the therapy.

ELIGIBILITY:
Inclusion Criteria

* Patients must have histologically or cytologically confirmed glioblastoma multiforme, anaplastic astrocytoma, or gliosarcoma.
* Prior therapy: Patients must have failed external beam radiotherapy to the brain, and if eligible and tolerated, undergone appropriate treatment with temozolomide chemotherapy. All radiation and additional chemotherapies must have been completed at least 4 weeks prior to enrollment. Prior therapy with nitrosoureas must have been completed at least 6 weeks prior to enrollment.
* Age ≥18 years (age of majority for clinical trials in Alabama). Because no dosing or adverse event data are currently available on the use of M032 in patients <18 years of age, children are excluded from this study but will be eligible for future pediatric phase 1 single-agent trials.
* Karnofsky Performance Status ≥70%
* Life expectancy of greater than 4 weeks.
* Patients must have normal organ and marrow function as defined below:

  * Leukocytes: >3,000/μl
  * absolute neutrophil count: >1,500/μl
  * platelets: >100,000/μl
  * total bilirubin within normal institutional limits
  * AST(SGOT)(aspartate aminotransferase)/ALT(SGPT)(alanine aminotransferase): <2.5 X institutional upper limit of normal
  * creatinine within normal institutional limits OR
  * creatinine clearance: >60 mL/min/1.73 m2 for patients with creatinine levels above institutional normal.
* Residual lesion must be ≥1.0 cm and < 5.5 cm in diameter without bilateral extension through the corpus callosum as determined by MRI as this is a locally delivered treatment. These parameters will be re-evaluated on imaging done on the day of catheter implantation and if the lesion no longer meets.
* The effects of M032 on the developing human fetus are unknown. For this reason, women of child-bearing potential and men must agree to use adequate contraception prior to study entry and for the first six months after receiving M032. Because it is currently unknown if M032 can be transmitted by sexual contact, a barrier method of birth control must be employed and for six (6) months following the administration of the study drug. Should a woman become pregnant while participating in this study, she should inform her treating physician immediately. For two weeks after receiving M032, subjects should avoid intimate contact with pregnant women, infants and young children and individuals with decreased immunity (ability to fight infection). Subjects should also refrain from donating blood during the trial
* Ability to understand and the willingness to sign a written informed consent document.
* Females of childbearing potential must not be pregnant; this will be confirmed by a negative serum pregnancy test within 14 days prior to starting study treatment.
* Steroid use is allowed as long as dose has not increased within 2 weeks of scheduled M032 administration. Whenever possible, the patient should be on a steroid dose that is equivalent to a dexamethasone dose of ≤ 2mg daily at the time of treatment.

Exclusion Criteria

* Patients who have had chemotherapy, cytotoxic therapy, immunotherapy within 4 weeks prior to entering the study (6 weeks for nitrosoureas), surgical resection within 4 weeks prior to entering the study, or have received experimental viral therapy or gene therapy at any time (e.g., adenovirus, retrovirus or herpes virus protocol). However, this does not preclude re-treatment with M032 at a later date.
* Patients who have not recovered from adverse events due to therapeutic interventions administered more than 4 weeks earlier.
* Patients may not be receiving any other investigational agents.
* History of allergic reactions attributed to compounds of similar biologic composition to M032 or to IL-12.
* Tumor involvement which would require ventricular, brainstem, basal ganglia, or posterior fossa inoculation or would require access through a ventricle in order to deliver treatment. Also, since M032 is a local treatment, patients whose tumors have bilateral extension through the corpus callosum, those with actively growing multifocal disease by MRI, and/or CSF dissemination/ leptomeningeal disease, are ineligible.
* Prior history of encephalitis, multiple sclerosis, or other CNS infection.
* Required steroid increase within 2 weeks of scheduled M032 administration. When possible, the patient should be on a dexamethasone equivalent dose of ≤ 2mg daily at the time of treatment.
* Active oral herpes lesion.
* Concurrent therapy with any drug active against HSV (acyclovir, valacyclovir, penciclovir, famciclovir, gancyclovir, foscarnet, cidofovir).
* Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or any other medical condition that precludes surgery. Also, psychiatric illness/social situations that would limit compliance with study requirements.
* Excluded patient groups

  * Pregnant women are excluded from this study because M032 is a viral oncolytic therapy with unknown potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with M032, breastfeeding women will not be included in the study.
  * Because patients with immune deficiency will be unable to mount the anticipated immune response underlying this therapeutic rationale, HIV-seropositive patients are excluded from this study. Other treatment studies for this disease that are less dependent on the patients' immune response are more appropriate for HIV-seropositive patients.
* Patients with known history of allergic reaction to IV contrast material that is not amenable to pre-treatment by University of Alabama at Birmingham protocol.
* Patients with pacemakers, ferro-magnetic aneurysm clips, metal infusion pumps, metal or shrapnel fragments or certain types of stents.
* Receipt of Gliadel Therapy.
* (Receipt of Bevacizumab (Avastin) therapy within 4 weeks of scheduled M032 administration. (Receipt of Bevacizumab (Avastin) greater than 4 weeks of scheduled M032 administration does not exclude patient.)
* Any other reason the investigator deems subject is unfit for participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2013-11-25 (Actual); Primary Completion 2022-09 (Actual); Study Completion 2027-09 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: James M. Markert, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- 10^5 Single Dose of HSV-1 (M032): Participants were administered 10^5 single dose of HSV-1 (M032) infused through catheters into region(s) of tumor defined by MRI
- 10^6 Single Dose of HSV-1 (M032): Participants were administered 10^6 single dose of HSV-1 (M032) infused through catheters into region(s) of tumor defined by MRI
- 10^7 Single Dose of HSV-1 (M032): Participants were administered 10^7 single dose of HSV-1 (M032) infused through catheters into region(s) of tumor defined by MRI
- 10^7.5 Single Dose of HSV-1 (M032): Participants were administered 10^7.5 single dose of HSV-1 (M032) infused through catheters into region(s) of tumor defined by MRI
- 10^8 Single Dose of HSV-1 (M032): Participants were administered 10^8 single dose of HSV-1 (M032) infused through catheters into region(s) of tumor defined by MRI
- 10^8.5 Single Dose of HSV-1 (M032): Participants were administered 10^8.5 single dose of HSV-1 (M032) infused through catheters into region(s) of tumor defined by MRI
- 10^9 Single Dose of HSV-1 (M032): Participants were administered 10^9 single dose of HSV-1 (M032) infused through catheters into region(s) of tumor defined by MRI
- Screen Fails: Participants that consented to the study, but ended up becoming ineligible before they were given M032
Period: Overall Study
Arm/Group | 10^5 Single Dose of HSV-1 (M032) | 10^6 Single Dose of HSV-1 (M032) | 10^7 Single Dose of HSV-1 (M032) | 10^7.5 Single Dose of HSV-1 (M032) | 10^8 Single Dose of HSV-1 (M032) | 10^8.5 Single Dose of HSV-1 (M032) | 10^9 Single Dose of HSV-1 (M032) | Screen Fails
Started | 4 | 1 | 1 | 2 | 6 | 1 | 6 | 8
Completed | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Not Completed | 4 | 1 | 1 | 2 | 6 | 0 | 5 | 8
Not completed — Death | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 3 | 1 | 1 | 2 | 6 | 0 | 5 | 0
Not completed — Screen Fail | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 8

BASELINE CHARACTERISTICS:
Groups:
- Screen Fails: Participants who consented, but became ineligible prior to receiving M032
- Total: Total of all reporting groups
Arm/Group | 10^5 Single Dose of HSV-1 (M032) | 10^6 Single Dose of HSV-1 (M032) | 10^7 Single Dose of HSV-1 (M032) | 10^7.5 Single Dose of HSV-1 (M032) | 10^8 Single Dose of HSV-1 (M032) | 10^8.5 Single Dose of HSV-1 (M032) | 10^9 Single Dose of HSV-1 (M032) | Screen Fails | Total
Number analyzed (Participants) | 4 | 1 | 1 | 2 | 6 | 1 | 6 | 8 | 29
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 4 | 1 | 1 | 2 | 5 | 1 | 5 | 7 | 26
  >=65 years | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 40 (48.45) | 39 (48.45) | 56 (48.45) | 42.5 (48.45) | 52.67 (48.45) | 56 (48.45) | 48.83 (48.45) | 50 (48.5) | 49.07 (48.45)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 1 | 0 | 1 | 1 | 0 | 2 | 7
  Male | 2 | 1 | 0 | 2 | 5 | 0 | 6 | 6 | 22
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 4 | 1 | 1 | 2 | 6 | 1 | 6 | 8 | 29
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 4 | 1 | 1 | 2 | 6 | 1 | 6 | 8 | 29

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD) of M032
Time Frame: baseline to12 months
Measure: Number; unit: plaque-forming units (PFU)
Groups:
- Single Dose of HSV-1 (M032): Participants were administered 10^5, 10^6, 10^7, 10^7.5, 10^8, 10^8.5, or 10^9 pfu of single dose of HSV-1 (M032) infused through catheters into region(s) of tumor defined by MRI
Arm/Group | Single Dose of HSV-1 (M032)
Number analyzed (Participants) | 21
plaque-forming units (PFU) | 1000000000

2. Secondary Outcome: Time to Progression Assessment
Time Frame: baseline to 12 months
Reporting Status: Not Posted

3. Secondary Outcome: The Time of Survival Assessment
Time Frame: baseline to 12 months
Reporting Status: Not Posted

4. Secondary Outcome: The Time of Biologic Assessment
Time Frame: baseline to 12 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | 10^5 Single Dose of HSV-1 (M032) | 10^6 Single Dose of HSV-1 (M032) | 10^7 Single Dose of HSV-1 (M032) | 10^7.5 Single Dose of HSV-1 (M032) | 10^8 Single Dose of HSV-1 (M032) | 10^8.5 Single Dose of HSV-1 (M032) | 10^9 Single Dose of HSV-1 (M032)
All-Cause Mortality (participants affected / at risk) | 4/4 | 1/1 | 1/1 | 2/2 | 6/6 | 1/1 | 4/6
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/1 | 0/1 | 1/2 | 1/6 | 1/1 | 2/6
Other Adverse Events (participants affected / at risk) | 4/4 | 0/1 | 0/1 | 2/2 | 6/6 | 1/1 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 10^5 Single Dose of HSV-1 (M032) (N=4) | 10^6 Single Dose of HSV-1 (M032) (N=1) | 10^7 Single Dose of HSV-1 (M032) (N=1) | 10^7.5 Single Dose of HSV-1 (M032) (N=2) | 10^8 Single Dose of HSV-1 (M032) (N=6) | 10^8.5 Single Dose of HSV-1 (M032) (N=1) | 10^9 Single Dose of HSV-1 (M032) (N=6)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cerebral Herniation (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Coma (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyponatremia (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Intracranial Infection - intradural (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Left Hemiplegia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea & vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory Insufficiency (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Right Lower Extremity Monoplegia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Strokes, bilateral (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Worsening Papular, Pustular rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Edema Left ankle/foot (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Surgical wound not healing (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 10^5 Single Dose of HSV-1 (M032) (N=4) | 10^6 Single Dose of HSV-1 (M032) (N=1) | 10^7 Single Dose of HSV-1 (M032) (N=1) | 10^7.5 Single Dose of HSV-1 (M032) (N=2) | 10^8 Single Dose of HSV-1 (M032) (N=6) | 10^8.5 Single Dose of HSV-1 (M032) (N=1) | 10^9 Single Dose of HSV-1 (M032) (N=6)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Aphasia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Ataxia (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bilateral nystagmus (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blurred Vision (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0
Body Aches (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bowel incontinence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bruising (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
BUE tremors (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Classic Candida Rash to groin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Constant black floaters (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Corneal abrasion (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chest Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Crush injury to right elbow (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Decreased fine motor movement (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Decreased visual field left eye, left side (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diplopia (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Dysesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ear Infection (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Elevated blood pressure (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Emesis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Enuresis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 3 (4) | 0 (0) | 2 (3)
Fecal incontinence (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fine motor slowing right hand (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gait Disturbance (Nervous system disorders) | 3 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypernatremia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Increased blood urea nitrogen (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Increased left sided weakness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Itching/dry eyes (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Itching/Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Left ankle sprain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Left arm & Right leg pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Left facial weakness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Left upper extremity weakness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0
Left eye double vision (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Left lower extremity muscle weakness against resistance (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Left lower extremity weakness (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Left side proprioception (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Left side weakness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lose of Balance (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Muscle weakness right side (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea & vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Non-pruritic red raised pustule rash on face, chest and back (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain & swelling L foot/ankle gout flare up (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Petechia left arm (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Psoriasis - worsening (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Right facial droop (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Right hip joint pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash to arms (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Redness to arms and legs (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Right hand weakness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Right lower extremity weakness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Right side eye and cheek swelling (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Right upper extremity weakness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Runny nose (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Sinus Congestion (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin discoloration red area back & abdomen (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sleepiness (General disorders) | 0 (0) | 0 | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Somnolence (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Sore throat (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Spasms (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tingling LLE (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary flow issues (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary Retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Quadrantanopia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Visual field deficit left (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Word finding difficulty (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Worsening balance, coordination and right side weakness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Worsening hemiparesis, left (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Yellow/Brown drainage left ear (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2023-08-10): https://cdn.clinicaltrials.gov/large-docs/27/NCT02062827/Prot_SAP_ICF_000.pdf